CLINICAL TRIAL: NCT06469905
Title: Effects of Erector Spina Plan Block and Exercise in Patients With Lumbar Disc Herniation
Brief Title: Erector Spina Plan Block in Patients With Lumbar Disc Herniation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Songül Bağlan Yentür, Head of Physiotherapy and Rehabilitation Department, Firat University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/06-39
Record Dates: First submitted 2024-06-14; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Low Back Pain
Keywords: Low back pain; Erector spina plane block; Exercise
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spina Plan Block group (Experimental): ESPB will be applied to the patients in the study group. Stabilization exercises will be applied together with ESPB treatment. The needle will be inserted between the erector spinae muscle and the transverse process structures.The local anesthetic will be monitored to spread along the erector spinae muscle.
  Interventions: Device: Erector Spina Plan Block; Other: Stabilization exercises
- Stabilization exercises group (Experimental): Stabilization exercises will be practiced to control group
  Interventions: Other: Stabilization exercises

INTERVENTIONS:
Device: Erector Spina Plan Block — ESPB will be applied to the patients in the study group. Stabilization exercises will be applied together with ESPB treatment. The needle will be inserted between the erector spinae muscle and the transverse process structures.The local anesthetic will be monitored to spread along the erector spinae muscle.
  Arms: Erector Spina Plan Block group
Other: Stabilization exercises — Stabilization exercises will be practiced to control group

SUMMARY:
Erector Spina Plan Block (ESPB) is a technique used in surgical interventions, acute and chronic pain. The aim of this study was to investigate the effect of ESPB and core stabilization exercises on functionality in patients with Lumbal Disc Herniation. ESPB will be applied to the patients in the study group. Stabilization exercises will be applied together with ESPB treatment. Only stabilization exercises will be applied to the patients in the control group. Patients will be asked to complete a questionnaire inquiring sociodemographic data (age, height, weight, BMI, smoking and alcohol use), VAS and Modified Oswestry Questionnaire at initial presentation and after 8 weeks of exercise (8 weeks 3 days a week).

DETAILED DESCRIPTION:
Low back pain is defined as pain in the lower back and/or legs that negatively affects comfort. Low back pain lasting less than 6 weeks is defined as acute, 6-12 weeks as subacute, and more than 12 weeks as chronic low back pain. The goals of the exercise program include reducing pain, strengthening weak muscles, stretching tense muscles, reducing mechanical stress on spinal structures, mobilizing hypomobile segments and stabilizing hypermobile segments. Erector Spina Plan Block (ESPB) is a technique used in surgical interventions, acute and chronic pain. The aim of this study was to investigate the effect of ESPB and core stabilization exercises on functionality in patients with Lumbal Disc Herniation. ESPB will be applied to the patients in the study group. Stabilization exercises will be applied together with ESPB treatment. The needle will be inserted between the erector spinae muscle and the transverse process structures.The local anesthetic will be monitored to spread along the erector spinae muscle. Only stabilization exercises will be applied to the patients in the control group. Patients will be asked to complete a questionnaire inquiring sociodemographic data (age, height, weight, BMI, smoking and alcohol use), VAS and Modified Oswestry Questionnaire at initial presentation and after 8 weeks of exercise (8 weeks 3 days a week).

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years old
* Patients diagnosed with disc herniation by clinical, physical examination and MR imaging
* Low back pain for >6 weeks

Exclusion Criteria:

* Severe spinal stenosis
* Diagnosis of pregnancy, infection or malignancy
* Presence of systemic inflammatory rheumatic disease
* Having neurological, orthopedic or congenital problems that prevent physical activity
* History of spinal surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2024-08-20 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
Disability assessment | 2 minutes
  Functional Disability Measurement; Assessment will be made using the Turkish version of the Modified Oswestry Questionnaire. n the evaluation of the Oswestry scale, the scoring for each question is A=0 B=1 C=2 D=3 E=4 F=5 points.

SECONDARY OUTCOMES:
Pain assessment | 1 minute
  Pain intensity will be assessed with a 10 cm Visuel Analog Scale (VAS). Patients are told what the numbers mean on the horizontal line, 0 means no pain, 10 means the most severe pain encountered in life, 5 means moderate pain and they are asked to describe the intensity of their pain on the scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Songul Baglan Yentur, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No